CLINICAL TRIAL: NCT01750632
Title: Subcapsular Orchiectomy in Men With Klinefelter Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: University of Copenhagen (Other); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jens Fedder, Professor, Consultant, Ph.D., Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lab.Reprod.Biol.-Horsens-02; M-20100041
Record Dates: First submitted 2012-12-08; First posted 2012-12-17 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Klinefelter Syndrome
MeSH Terms: conditions — Klinefelter Syndrome | interventions — Orchiectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Orchiectomy (Experimental): The patients undergo subcapsular orchiectomy
  Interventions: Procedure: Orchiectomy

INTERVENTIONS:
Procedure: Orchiectomy — The patients undergo subcapsular orchiectomy with basic surgical instruments. The patients are given local analgesia and sometimes universal anesthesia.

SUMMARY:
Men with Klinefelter syndrome undergo unilateral subcapsular ochiectomy, and the removed testicular tissue is examined for presence of sperm and cryopreserved in small pieces for fertility treatment and scientific purposes. Prior to operation blood samples are frozen in a biobank.

ELIGIBILITY:
Inclusion Criteria:

* Klinefelter
* 15-40 years of age

Exclusion Criteria:

* inability to understand the study

Ages: 15 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2010-08; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Presence of testicular sperm | Between 1 and 6 months

SECONDARY OUTCOMES:
Clinical pregnancy rate after ICSI with retrieved testicular sperm | participants will be followed for the duration of fertility treatment, an expected average of 6 months

OTHER OUTCOMES:
Predictive value of FSH and other hormones for the presence of testicular sperm | Between 1 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic, Odense University Hospital, Odense, Denmark

REFERENCES:
- [Result] Fedder J, Gravholt CH, Kristensen SG, Marcussen N, Engvad B, Milton AM, Andersen CY. Testicular Sperm Sampling by Subcapsular Orchiectomy in Klinefelter Patients: A New Simplified Treatment Approach. Urology. 2015 Oct;86(4):744-50. doi: 10.1016/j.urology.2015.06.044. Epub 2015 Aug 4. PMID 26254174